CLINICAL TRIAL: NCT04124263
Title: Use of Short Text Messages to Promote Medication Adherence in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Collaborators: Medtronic Foundation (Unknown)
Responsible Party: Principal Investigator, Márcio Galvão Guimarães de Oliveira, Adjunct Professor, Federal University of Bahia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 332/2016
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Hypertension; Adherence, Treatment
Keywords: Hypertension; Primary Health Care
MeSH Terms: conditions — Hypertension; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication Time Short Messages (Experimental): 70 hypertensive patients registered for access to medications that will additionally receive text messages at the times indicated in the prescription for use of each indicated medication, in addition to educational information.
  Interventions: Other: Educational short message texts; Other: Adherence short message texts
- Educational Short Messages (Experimental): 70 hypertensive patients registered for access to medications that will additionally receive text messages at the times indicated in the prescription for use of each indicated medication, in addition to educational information.
  Interventions: Other: Educational short message texts; Other: Adherence short message texts

INTERVENTIONS:
Other: Educational short message texts — Educational messages for patient engagement
Other: Adherence short message texts — Reminder messages of medication use time

SUMMARY:
OBJECTIVE: To evaluate the effect of intervention by sending short text messages with a reminder of the time of medication use, compared to sending educational messages, on adherence to drug treatment in patients with hypertension. METHODOLOGY: Prospective, randomized, controlled, double-blind, parallel group study that will be performed in patients with hypertension seen at a community pharmacy in Brazil. The following groups will be compared: a) intervention group 1: 70 hypertensive patients registered for access to medication associated with usual care, in addition to text messages via mobile phone with educational information b) intervention group 2: 70 hypertensive patients registered for access to medications that will additionally receive text messages at the times indicated in the prescription for use of each indicated medication, in addition to educational information. After the washout period, the groups will have the active interventions changed for an additional 90 days. The proportion of adherent and non-adherent patients with and without controlled BP in both groups will be compared after the periods of application of the different interventions.

ELIGIBILITY:
Inclusion Criteria: hypertension diagnosis, age, availability of mobile phone with short message texts access and ability to read and access short message texts -

Exclusion Criteria: visual, hearing or mental disabilities that disables receiving short message texts , being pregnant, recently delivered or breastfeeding

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Treatment adherence | Seven months (including one month of washout period)
  Measurement of medication usage through Brief Medication Questionnaire: low to high adherence

SECONDARY OUTCOMES:
Blood pressure | Seven months (including one month of washout period)
  Measurement of blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Farmácia Escola da UFBA, campus Anísio Teixeira, Vitória da Conquista, Estado de Bahia, Brazil